CLINICAL TRIAL: NCT02814383
Title: Diastolic Closing Margin Predicts Brain Injury in Premature Infants
Brief Title: Prediction of Brain Injury in Premature Infants
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Christopher J. Rhee, MD, MS, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-38084; K23NS091382 (NIH)
Record Dates: First submitted 2016-05-26; First posted 2016-06-27 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Intraventricular Hemorrhage; Periventricular Leukomalacia; Brain Injury; Extreme Prematurity
Keywords: Prematurity; Extremely Low Birth Weight (ELBW); Cerebral Perfusion; Cerebral Autoregulation
MeSH Terms: conditions — Leukomalacia, Periventricular; Brain Injuries; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ELBW Infants: This study seeks to collect data on premature ELBW infants (less than or equal to 2.2 lbs) at high risk of developing brain injury.
  Interventions: Other: Brain Monitoring Platform

INTERVENTIONS:
Other: Brain Monitoring Platform — This study is being done to evaluate the changes in brain perfusion measured by the DCM using a comprehensive and innovative brain monitoring platform that encompasses direct and continuous measures of cerebral blood flow (CBF), cerebral oximetry, cerebral autoregulation, partial pressure of carbon dioxide (PCO2), and arterial blood pressure (ABP).

SUMMARY:
Extremely low birth weight (ELBW), birth weight less than or equal to 1000 g, infants are at high risk for developing brain injury in the first week of life. Intraventricular hemorrhage (IVH) and periventricular leukomalacia (PVL) are the most common injuries in this group of infants. Their incidence is inversely proportional to gestational age (GA) and birth weight (BW). These lesions are associated with neurodevelopmental delay, poor cognitive performance, visual and hearing impairment, epilepsy, and cerebral palsy; and instability of systemic hemodynamics during transition from intra- to extra-uterine life and during the early neonatal period is believed to be at their genesis. While the incidence of ultrasound- diagnosed cystic PVL has decreased dramatically over the last 2 decades, diffuse PVL detected by magnetic resonance imaging (MRI) is still prevalent in survivors of neonatal intensive care. Moreover, PVL, even when non-cystic, is associated with decreased cortical complexity and brain volume and eventual neurocognitive impairment.

Currently, clinicians lack the tools to detect changes in cerebral perfusion prior to irreversible injury. Unfortunately, the incidence of brain injury in ELBW infants has remained relatively stable. Once translated to the bedside, the goal of this research is to develop a monitoring system that will allow researchers to identify infants most at risk for IVH and PVL and in the future, intervention studies will be initiated to use the changes in cerebral perfusion to direct hemodynamic management.

The purpose of this study is to first understand the physiology of brain injury and then to eventually impact the outcomes in this high-risk group of infants by assessing the ability of the diastolic closing margin (DCM), a non-invasive estimate of brain perfusion pressure, to predict hemorrhagic and ischemic brain injury in ELBW infants. The information collected for this study will help develop algorithms or monitoring plans that will maintain the appropriate brain perfusion pressure and thereby, prevent severe brain injury.

DETAILED DESCRIPTION:
This is a prospective, single-center, data collection research study for premature ELBW infants at high risk of developing brain injury. This study is being done to evaluate the changes in brain perfusion measured by the DCM using a comprehensive and innovative brain monitoring platform that encompasses direct and continuous measures of cerebral blood flow (CBF), cerebral oximetry, cerebral autoregulation, partial pressure of carbon dioxide (PCO2), and arterial blood pressure (ABP) in the hopes to both describe the physiology of brain injury and to correlate these findings to short- and long-term outcomes relevant to ELBW infants.

About three hundred and ten (310) subjects are expected to be enrolled. Subjects' active participation in the study may last up to one week and the total time they will be followed after birth is approximately 24 months (2 years) or more (+/- 2 Months) depending on their prematurity. Information from the subjects' medical records may be accessed, reviewed, and recorded for an additional year after their final study visit. This study consists of about 5 study visits: Study Visit 1 (the enrollment visit - within first 12 hours of life), Study Visit 2 (occurs 2-7 days post visit 1), Study Visit 3 (occurs approximately 2-4 months +/- 2 Months term equivalent age/corrected age of the subject ), Study Visit 4 (occurs approximately at 12 months +/- 2 Months corrected age of the subject), and Study Visit 5 (occurs approximately at 18-24 months +/- 2 Months chronological age of the subject).

STUDY ASSESSMENTS:

* Medical and Surgical History: The subjects' detailed history will be reviewed and recorded. The subjects' mothers will also be asked questions about their own medical history. The mothers' medical records may also be accessed.
* Continuous Physiologic Monitoring: Monitoring will be performed that includes the transcranial Doppler ultrasound, near-infrared spectroscopy (NIRS), and partial pressure of carbon dioxide (PCO2) from birth to 7 days of life (visits 1 and 2).
* Ventilator: The highest daily ventilator settings and mean airway pressure (MAP) will be reviewed and recorded from birth to 7 days of life (visits 1 and 2).
* Head Ultrasound: A head ultrasound will be performed upon enrollment (visit 1) to assess for early and preexisting brain injury (IVH).
* Adverse Events: Any adverse events (AEs), special events of interest, or unanticipated problems (UPs) that subjects may have experienced after enrollment will be reviewed and recorded (visits 1, 2, 3, 4, and 5).
* Concomitant Medications: Review and record any medications of interest that subjects are taking from birth to 7 days of life (visits 1 and 2).
* Blood Transfusions: Review and record the transfusion of blood products that are performed on the subjects as part of standard of care from birth to 7 days of life (visits 1 and 2).
* Echocardiogram (ECG) and Head Ultrasound: Review and record ECG and head ultrasound results that are performed on the subjects as part of standard of care from birth to 7 days of life (visits 1 and 2).
* Respiratory Interventions and Suctioning: Review and record any respiratory interventions and/or suctioning that are performed on the subjects as part of standard of care from birth to 7 days of life (visits 1 and 2).
* Magnetic Resonance Imaging (MRI): Perform a MRI exam at visit 3 or up to the time of discharge.
* Capute Scales and Neurologic Exam: Perform this assessment at visit 4 to assess the subjects' development and cognitive function and to provide an early evaluation for any neurologic abnormalities that may be related to brain injury.
* Bayley-III Motor Sub-Test Exam: Perform this assessment at visit 4 to assess the subjects' development and cognitive function and to provide an early evaluation for any neurologic abnormalities that may be related to brain injury.
* Complete Bayley-III Exam: Perform this assessment at visit 5 to assess the subjects' development and cognitive function and to provide an early evaluation for any neurologic abnormalities that may be related to brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from parent or legally authorized representative (LAR)
* Live-born ELBW infant
* Less than 12 hours of life
* Birth weight 401 to 1000g
* Admitted to Texas Children's Hospital (TCH) Pavilion for Women (PFW) Neonatal Intensive Care Unit (NICU)
* Umbilical arterial catheter (UAC) in place

Exclusion Criteria:

* Complex congenital anomalies of central nervous system (CNS)
* Complex chromosomal congenital anomalies
* Hydrops fetalis
* Poor skin integrity
* Live-born but receiving only comfort care
* Grade 3-4 IVH by head ultrasound (HUS) at the first ultrasound completed at or before 12 hours of life

Ages: 0 Hours to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Within 12 hours of life, subjects' mothers will be approached for participation in this research study. This study seeks to collect data on premature ELBW infants (less than or equal to 2.2 lbs) at high risk of developing brain injury.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2016-08-11 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Brain Perfusion | 1 Week
  Brain perfusion will be assessed by calculating the diastolic closing margin (DCM). DCM will be measured from continuous recordings of middle cerebral artery cerebral blood flow velocity (CBFV) by transcranial Doppler ultrasound and ABP during first week of life for ELBW infants.

SECONDARY OUTCOMES:
Brain Perfusion | 1 Week
  Brain perfusion will be assessed by calculating the systolic blood flow autoregulation.
Brain Perfusion | 1 Week
  Brain perfusion will be assessed by calculating the critical closing pressure (CrCP).
Brain Injury (IVH) | 1 Week
  The presence of IVH will be assessed by two head ultrasounds (HUS).
Brain Injury (PVL) | 7 Weeks
  The presence of PVL will be assessed by magnetic resonance imaging (MRI) at term-equivalent age (date on which patient reaches 37 to 40 weeks post-conception age) using conventional MRI.
Brain Injury (PVL) | 7 Weeks
  The presence of PVL will be assessed by magnetic resonance imaging (MRI) at term-equivalent age (date on which patient reaches 37 to 40 weeks post-conception age) using quantitative diffusion tensor imaging.
Neurodevelopmental Function | 12 Months
  Neurodevelopmental function will be assessed using the Bayley III motor subtest at 12 months.
Neurodevelopmental Function | 12 Months
  Neurodevelopmental function will be assessed using the neurologic exam at 12 months.
Neurodevelopmental Function | 12 Months
  Neurodevelopmental function will be assessed using the Capute Scales at 12 months.
Neurodevelopmental Function | 24 Months
  Neurodevelopmental function will be assessed using the Bayley III motor subtest at 18-24 Months.
Neurodevelopmental Function | 24 Months
  Neurodevelopmental function will be assessed using the Bayley III language subtest at 18-24 Months.
Neurodevelopmental Function | 24 Months
  Neurodevelopmental function will be assessed using the Bayley III cognitive subtest at 18-24 Months.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J. Rhee, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Baylor College of Medicine, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Texas Children's Pavilion for Women, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description Dr. Rhee's Profile Page — https://www.texaschildrens.org/find-a-provider/christopher-j-rhee-md-ms